CLINICAL TRIAL: NCT03340324
Title: Open Label, One-arm, 2-month Study of Once-daily Tablet of V-Endo as Immunotherapy of Endometriosis
Brief Title: Open Label Immunotherapy of Endometriosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Collaborators: Ekomed LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-Endo
Record Dates: First submitted 2017-10-11; First posted 2017-11-13 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Endometriosis
Keywords: inflammation; autoimmunity; immunotherapy; infertility; pelvic pain
MeSH Terms: conditions — Endometriosis; Inflammation; Autoimmune Diseases; Infertility; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: open-label, single arm study
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm open label V-Endo recepients (Experimental): This is single arm open label trial wherein active drug is V-Endo
  Interventions: Biological: V-Endo

INTERVENTIONS:
Biological: V-Endo — V-Endo is a tableted immunotherapeutic derived from hydrolyzed, heat-inactivated, pooled blood from women with endometriosis

SUMMARY:
Endometriosis is a chronic gynecological disease characterized by sustained painful symptoms that are responsible for a decline in the quality of life of sufferers. Endometriosis is fairly common, affecting an estimated 10%-15% of women and girls, usually during their reproductive years. Based on these rough estimates, the latest epidemiological studies suggest that over 200 million women are might be affected who may commonly have infertility problems. Additionally, endometriosis is a major factor increasing by 33-66% risk of ovarian cancer. V-Endo is a tableted preparation derived from hydrolyzed, heat-inactivated, pooled blood of women with endometriosis. When taken orally it is postulated to cause the immune tolerance and anti-inflammatory effect as a result.

DETAILED DESCRIPTION:
Anatomically endometriosis is characterized by the presence of endometrial-type mucosa outside the uterine cavity. This tissue proliferates and causes chronic inflammation resulting in pain and excessive menstrual bleeding. Conventional treatment includes surgical and pharmacological therapy aiming at reducing painful symptoms. However, there is an unmet need in finding optimally safe and effective treatment. This study aimed to evaluate the effect of V-Endo on pain levels in women with endometriosis, focusing on reducing inflammation by immunotherapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years
* pain visual analog scale (VAS) score over 4 (visual linear scale from 0 to 10)
* confirmation of endometriosis by laparoscopy
* no drugs used at least for one month prior to enrollment, i.e., estro-progestinic, progestinic, gonadotropin-releasing hormone (GnRH) agonists and antagonists as well as nonsteroidal anti-inflammatory drugs (NSAIDs)

Exclusion Criteria:

* presence of other associated diseases such as malignancies
* concomitant use of hormonal drugs
* menopause
* pregnancy
* surgery for endometriosis within the last month prior to study entry
* unable or unwilling to give written consent patients
* adverse reaction or hypersensitivity to active substance or excipients of V-Endo

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females will be enrolled as only they have endometriosis
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect on pelvic pain by visual analogue scale (VAS) | 2 months
  The pain VAS is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).

SECONDARY OUTCOMES:
Effect of V-Endo on complete blood count (CBC) | 2 months
  The effect of V-Endo on complete blood cell count and clinical biochemistry will be evaluated by routine lab tests to determine whether they are within normal ranges are as described in http://onlinelibrary.wiley.com/doi/10.1002/9781118704783.app3/pdf
Changes induced By V-Endo on life quality | 2 months
  Changes in life quality occurring as a result of intervention as measured by EHP-30 instrument https://innovation.ox.ac.uk/outcome-measures/endometriosis-health-profile-ehp/
Effect of V-Endo liver and kidney biochemistry parameters | 2 months
  The influence on kidney and liver biochemistry parameters measured as described in http://onlinelibrary.wiley.com/doi/10.1002/9781118704783.app3/pdf

CONTACTS AND LOCATIONS:
Overall Officials: aldar bourinbaiar, MD/PhD, Study Chair — CEO
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: Undecided
Once trial is terminated data will be available to share